CLINICAL TRIAL: NCT06761274
Title: Study of Epigenetic and Inflammatory Markers of Accelerated Biological Ageing in the Follow-up of Patients With Hodgkin's Lymphoma in Complete Remission for at Least 2 Years
Brief Title: Study of Epigenetic and Inflammatory Markers of Accelerated Biological Ageing in the Follow up of Patients With Hodgkin's Lymphoma
Acronym: MEPI-AGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MEPI-AGE; PR 1/CS/AIL/21 (Other Grant/Funding Number: AIL Bologna ODV); RC-2022-2773333 (Other Grant/Funding Number: Ricerca Corrente 2022-2024 (Ministero della Salute))
Record Dates: First submitted 2024-12-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Hodgkin Lymphoma in Remission
Keywords: epigenetic markers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hodgkin lymphoma patients in complete remission for at least two years and newly diagnosed (Experimental): in vitro human tissue testing of peripheral blood in hodgkin lymphoma patients in complete remission for at least two years after first-line therapy with stage II b, III or IV
  Interventions: Other: peripheral blood sampling

INTERVENTIONS:
Other: peripheral blood sampling — It is a monocentric and exploratory study, experimental on human tissues in vitro and similar projects do not exist in the literature. This study involves the analysis of peripheral blood in patients with hodgkin lymphoma with the following characteristics:
  * in complete remission for at least two years after first-line therapy with stage II b, III or IV at onset (Ann Arbor classification).
  * newly diagnosed (stage II b, III or IV, Ann Arbor Classification).

SUMMARY:
Study design: It is a monocentric and exploratory study, experimental on human tissues in vitro which involves the analysis of peripheral blood in patients with Hodgkin's lymphomas with the following characteristics:

* in complete remission for at least two years after first-line therapy with stage IIb, III or IV at onset (Ann Arbor classification).
* newly diagnosed (stage IIb, III or IV, Ann Arbor Classification).

DETAILED DESCRIPTION:
The study aims to evaluate patients with hodgkin lymphoma in complete remission for at least 2 years and newly diagnosed (stage II b, stage III or stage IV) as they are currently characterised by a long life expectancy during which there is an increased and early incidence of non-neoplastic systemic complications as well as, of course, manifestations of secondary malignancies.

ELIGIBILITY:
Inclusion Criteria:

* hodgkin lymphoma stage II b, III or IV at onset in remission for at least two years after the first line of therapy for lymphoma
* Newly diagnosed histologically confirmed stage II b, III or IV patients who require first-line therapy
* Patients of both sexes aged ≥ 18 years at enrollment
* Signature of informed consent

Exclusion Criteria:

* Concomitant second neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
evaluation of senescence markers (CD57, KLRG1,CD62L, CD45RA) | through study completion, an average of 2 year
  Determine the biological age of patients
DNA methylation (methylation rate) | through study completion, an average of 2 year
  Determine the biological age of patients

SECONDARY OUTCOMES:
evaluation of senescence markers (CD57, KLRG1,CD62L, CD45RA) | through study completion, an average of 2 year
  Determine the possible acceleration of the biological age of patients
DNA methylation (methylation rate) | through study completion, an average of 2 year
  Determine the possible acceleration of the biological age of patients

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No